CLINICAL TRIAL: NCT05762978
Title: Negative Inspiratory Flow (NIF) in Children Age 4-8 Years During Acute Asthma to Evaluate the Use of a Dry Powder Inhaler: A Pilot Study
Brief Title: Evaluation of Negative Inspiratory Flow in Children With Acute Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15035
Record Dates: First submitted 2016-04-14; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthmatic Children (Experimental): NIF will be measured using an In-Check Dial
  Interventions: Device: In-Check Dial; Device: Inhaler Device

INTERVENTIONS:
Device: In-Check Dial — Patient will have their NIF measured with In-Check Dial
Device: Inhaler Device — Children will use inhaler per standard of care.

SUMMARY:
There are different inhalers used for the treatment of asthma and they work differently and require different technique for the optimal drug delivery to the lungs. One of the inhalers is the Dry Powder Inhaler (DPI). The minimal amount of Negative Inspiratory Flow (NIF) required to use this medication is 30ml/min. Studies have shown that children find it difficult to generate this NIF and studies have also shown that children generate lesser NIF during an Asthma exacerbation. The investigators will measure the NIF using an InCheck Dial on children with asthma during an exacerbation and when they are seen in clinic for a hospital follow up visit. This will be done on asthmatic children regardless of the inhaler that they use. The investigator hypothesize that children with asthma age 4-8 years cannot generate the required NIF during an Asthma exacerbation hence proving that a DPI cannot be prescribed to children at this age. This study will examine this hypothesis.

DETAILED DESCRIPTION:
Inhaler devices are the major method for delivery of asthma medication, but their effectiveness can be compromised if the patient uses the inhaler device incorrectly. The magnitude of this problem has been well documented; in several studies less than half of the patients used their inhaler correctly. Inhaler devices are used to deliver a variety of inhaled medications, including beta-agonists, anticholinergic, and glucocorticoids. Two main types of inhaler devices are available, the pressurized metered dose inhaler (pMDI) and the dry powder inhaler (DPI).

A dry powder inhaler (DPI) is a breath-actuated device containing micronized drug particles with a mass median aerodynamic diameter (MMAD) of less than 5 µm that are usually aggregated with carrier particles (such as lactose or glucose) of greater diameter. Drug is delivered to the airways by the inhalation of air over a punctured drug-containing capsule or blister.

In this study investigators will evaluate the use of DPI use in children during an acute asthma exacerbation. The investigators hypothesize the use of DPI in children ages 4-8 during an asthma exacerbation has limited benefit, as children are unable to generate the needed NIF. The investigators will study children who were hospitalized for an acute asthma exacerbation. Additionally, the investigators will evaluate the participant as an outpatient in the pulmonary clinic / office when the participant is without an asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with asthma
* Age ≥ 4 years and < 8 years

Exclusion Criteria:

* Acute Lung Disease
* Chronic lung disease
* Developmental Delay

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2015-12; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
NIF (Negative Inspiratory Flow) | Time of Hospital Admission (Day 1)
  NIF measures a patient's maximum inspiratory effort after exhaling.
NIF (Negative Inspiratory Flow) | Hospital Discharge (Typically Day 1-2)
  NIF measures a patient's maximum inspiratory effort after exhaling.
NIF (Negative Inspiratory Flow) | Follow-Up Visits (Week 2 Post-Discharge)
  NIF measures a patient's maximum inspiratory effort after exhaling.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Halaby, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States